CLINICAL TRIAL: NCT03446651
Title: Mechanism and Effects of Manipulating Chloride Homeostasis in Acute Heart Failure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2000022001; 1R01HL139629-01 (NIH)
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
Keywords: Sodium Homeostasis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lysine Chloride (Experimental): Participants will be randomized to 7 days of therapy with either 115 mmol/day of lysine chloride or placebo. People in the Lysine Chloride group will receive the active intervention.
  Interventions: Drug: Lysine Chloride
- Placebo (Placebo Comparator): Participants will be randomized to 7 days of therapy with either 115 mmol/day of lysine chloride or placebo. People in the Placebo group will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lysine Chloride — Patients will receive 7 days of therapy using 115 mmol/day of lysine chloride. Patients will be given the option of a taste test of both lysine chloride & the placebo powders mixed with various beverages to ensure it is palatable to them. If the patient feels they will not be able to take the study medication twice a day due to taste, they will be withdrawn from the study at this time.
  Arms: Lysine Chloride
Other: Placebo — Patients will receive 7 days of therapy using placebo. Patients will be given the option of a taste test of both lysine chloride & the placebo powders mixed with various beverages to ensure it is palatable to them. If the patient feels they will not be able to take the study medication twice a day due to taste, they will be withdrawn from the study at this time.
  Arms: Placebo

SUMMARY:
The purpose of this study is to understand the effects of chloride supplementation on volume-overloaded acute heart failure patients concomitantly treated with IV diuretics.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to develop a comprehensive understanding of the biology and therapeutic potential of sodium-free chloride supplementation. While sodium homeostasis has been the focus of substantial investigation, very little research has been devoted to understanding chloride homeostasis. Thus, this proposal is designed to obtain the full spectrum of information pertaining to chloride, such as novel areas with great interest by the scientific community (i.e. modulation of the WNK-kinase system and the use of exosomes), to more practical/basic questions (i.e. what happens to sodium chloride balance when a patient is challenged with chloride). The proposed outpatient study has been designed to serve as a real world efficacy study. With extensive biobanking and analysis of samples in the proposed setting, there is the potential to be able to deliver a great wealth of information on the biology and therapeutic potential of manipulating chloride homeostasis in heart failure.

Research confirms that many heart failure therapies demonstrate measurable benefit in highly controlled environments, but lack effectiveness when studied in decompensated patients receiving standard decongestive therapies. As such, this study seeks to understand the effects of chloride supplementation on volume-overloaded patients concomitantly treated with IV diuretics.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of decompensated heart failure with at least one objective sign of volume overload (rales, edema, elevated jugular venous pressure (JVP), or weight gain of at least 5 pounds)
* A projected need by the treating clinician for continued treatment with IV diuretics
* Chronic loop diuretic use

Exclusion Criteria:

* Inability to commit to or comply with serial visits for treatment in the Yale Transitional Care Center (YTCC)
* History of severe metabolic or respiratory acidosis within 30 days of enrollment
* Use of metformin, acetazolamide, or any other agent that could predispose to acidosis. Patients who are on metformin may be enrolled if their metformin can be discontinued safely for the duration of the study. Any participants who have consistently elevated Blood glucose readings > 200 mg/dL while inpatient will not be enrolled.
* Serum bicarbonate level <20mmol/L
* Estimated glomerular filtration rate <20 mL/min or renal replacement therapy
* Appears unlikely, or unable to participate in the required study procedures, as assessed by the study PI or research registered nurse (RN) (ex: clinically-significant psychiatric, addictive, or neurological disease)
* Inability to give written informed consent or follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kazory A. Combination Diuretic Therapy to Counter Renal Sodium Avidity in Acute Heart Failure: Trials and Tribulations. Clin J Am Soc Nephrol. 2023 Oct 1;18(10):1372-1381. doi: 10.2215/CJN.0000000000000188. Epub 2023 Apr 27. PMID 37102974

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lysine Chloride | Placebo
Started | 22 | 18
Participated in Open Label Portion | 5 | 0
Completed 1st Visit | 17 | 18
Completed Final Visit | 13 | 18
Completed | 13 | 18
Not Completed | 9 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Open Label Participants | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lysine Chloride | Placebo | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.61) | 58.61 (13.68) | 56.30 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 16 | 13 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 11 | 8 | 19
  Race: Black | 10 | 8 | 18
  Race: Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 40
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 120.32 (24.66) | 129.44 (28.03) | 124.43 (26.28)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 71.59 (10.82) | 78.0 (15.43) | 74.47 (13.31)
Heart rate [Mean (Standard Deviation); unit: bpm] | 80.27 (16.93) | 88.11 (21.61) | 83.80 (19.33)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Volume
Description: Volumex is albumin labeled with the iodine isotope I-131 and is an FDA-approved method used to determine total blood volume. A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of blood collection will be compared across the 7 day collection period between intervention and placebo arms.
Time Frame: Daily for 7 days
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Lysine Chloride | Placebo
Number analyzed (Participants) | 22 | 18
mL | -320 (689) | -447 (520)
Statistical Analysis 1: Comparison: Lysine Chloride vs Placebo; Test type: Superiority; p = 0.56, t-test, 2 sided

2. Secondary Outcome: Change in Log NTpro-BNP
Description: N-terminal prohormone of brain natriuretic peptide (NTpro-BNP) is used to screen and diagnosis of acute congestive heart failure (CHF) and can be used to establish prognosis in heart failure. A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of NTpro-BNP will be compared across the 7 day collection period between intervention and placebo arms.
Time Frame: Daily for 7-days
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Change in Serum Creatinine
Description: A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of serum creatinine will be compared across the 7 day collection period between intervention and placebo arms.
Time Frame: Daily for 7-days
Population: Intention to treat
Measure: Mean (95% Confidence Interval); unit: mg/dL per day
Arm/Group | Lysine Chloride | Placebo
Number analyzed (Participants) | 22 | 18
mg/dL per day | 0.00 [-0.04 to 0.04] | 0.04 [0.02 to 0.06]
Statistical Analysis 1: Comparison: Lysine Chloride vs Placebo; Test type: Superiority; p = 0.039, t-test, 2 sided

4. Secondary Outcome: Change in Cystatin C
Description: A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of cystatin C will be compared across the 7 day collection period between intervention and placebo arms.
Time Frame: Daily for 7-days
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Change in Chloride
Description: A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of chloride will be compared across the 7 day collection period between intervention and placebo arms.
Time Frame: Daily for 7-days
Population: Intention to treat
Measure: Mean (95% Confidence Interval); unit: mmol/L per day
Arm/Group | Lysine Chloride | Placebo
Number analyzed (Participants) | 22 | 18
mmol/L per day | 0.71 [0.36 to 1.06] | -0.87 [-1.32 to -0.43]
Statistical Analysis 1: Comparison: Lysine Chloride vs Placebo; Test type: Superiority; p < 0.001, t-test, 2 sided

6. Secondary Outcome: Change in Bicarbonate
Description: A linear mixed effect model will be used to analyze the trial with class variables of time and treatment group. Daily measures of bicarbonate will be compared across the 7 day collection period between intervention and placebo arms.
Time Frame: Daily for 7-days
Population: Intention to treat
Measure: Mean (95% Confidence Interval); unit: mmol/L per day
Arm/Group | Lysine Chloride | Placebo
Number analyzed (Participants) | 22 | 18
mmol/L per day | -1.02 [-1.35 to -0.70] | 0.19 [-0.16 to 0.55]
Statistical Analysis 1: Comparison: Lysine Chloride vs Placebo; Test type: Superiority; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 7 days
Arm/Group | Lysine Chloride | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 12/22 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lysine Chloride (N=22) | Placebo (N=18)
Diarrhea (Gastrointestinal disorders) | 8 | 2
Renal failure (Renal and urinary disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Metabolic acidosis without acidemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
GI bloating (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gout (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This is preliminary data analysis conducted solely for the purpose of complying with clinicaltrials.gov timelines

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT03446651/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03446651/ICF_001.pdf